CLINICAL TRIAL: NCT07272226
Title: Comparison of the Effectiveness of Lumbar Plexus Block and Hypobaric Unilateral Spinal Anesthesia in Patients Undergoing Femoral Neck Fracture Surgery
Brief Title: Comparison of Unilateral Spinal Anesthesia and Nerve Block in Hip Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gokberk Kursat Ulker, Anesthesiology and Reanimation Resident, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011- KAEK-25 2023/07-14
Record Dates: First submitted 2025-01-06; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Femur Neck Fracture; Spinal Anesthesia; Lumbar Plexus Nerve Block
Keywords: Spinal Anesthesia; Lumbar Plexus Block; Femoral Neck Fracture; Regional Anesthesia; Peripheral Nerve Block
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hipobaric Unilateral Spinal Anesthesia Group (Experimental)
  Interventions: Procedure: Hipobaric Unilateral Spinal Anesthesia Group
- Lomber Plexus Block Group (Experimental)
  Interventions: Procedure: Lumbar Plexus Block (LP-SP)

INTERVENTIONS:
Procedure: Hipobaric Unilateral Spinal Anesthesia Group — Patients in this group receive hypobaric unilateral spinal anesthesia (HUSA) using 5 mg of 0.5% bupivacaine diluted with 3 mL of distilled water. The injection is administered at the L4-L5 intervertebral space in the lateral position. Hemodynamic parameters, sensory block levels, and intraoperative requirements are monitored.
  Arms: Hipobaric Unilateral Spinal Anesthesia Group
Procedure: Lumbar Plexus Block (LP-SP) — Patients in this group undergo lumbar plexus block (LP-SP) using a Shamrock or paramedian sagittal ultrasound-guided approach. A mixture of 0.5% bupivacaine and saline (total volume: 25-35 mL) is administered based on patient body weight (max 2.5 mg/kg). Neurostimulation is used to confirm accurate needle placement in the psoas muscle. Hemodynamic stability, block efficacy, and sedation needs are assessed.
  Arms: Lomber Plexus Block Group

SUMMARY:
This randomized study aims to compare the efficacy and hemodynamic effects of hypobaric unilateral spinal anesthesia (HUSA) and lumbar plexus block (LP-SP) in patients undergoing femoral neck fracture surgery. Conducted at a single center, the study includes 60 patients aged 18 to 90, classified as ASA I-IV, and evaluates anesthesia methods' impact on intraoperative parameters, including blood pressure, sedation needs, and recovery outcomes. The findings will inform anesthetic strategy selection based on patient characteristics and surgical requirements.

DETAILED DESCRIPTION:
This prospective, randomized, controlled study is designed to compare hypobaric unilateral spinal anesthesia (HUSA) and lumbar plexus block combined with sacral plexus block (LP-SP) in patients undergoing femoral neck fracture surgery. The study will be conducted at Bursa Yüksek İhtisas Training and Research Hospital and will include a total of 60 patients aged between 18 and 90 years with ASA physical status I-IV.

Eligible patients will be randomized into two groups: the HUSA group and the LP-SP group. In the HUSA group, unilateral spinal anesthesia will be performed using 5 mg of 0.5% bupivacaine diluted with distilled water to achieve a hypobaric solution. In the LP-SP group, lumbar plexus block and sacral plexus block will be performed using ultrasound-guided Shamrock or paramedian sagittal approaches with 0.5% bupivacaine.

Standard intraoperative monitoring will be applied to all patients, including electrocardiography, non-invasive blood pressure, pulse oximetry, and anesthesia depth monitoring with entropy and surgical pleth index. Intraoperative sedation, vasopressor use, and intravenous fluid administration will be managed according to institutional clinical protocols and patient needs.

Hemodynamic parameters, anesthesia depth indices, nociception indices, sedation requirements, and recovery-related parameters will be recorded intraoperatively at predefined time points. All data will be collected prospectively and analyzed to compare the two anesthetic techniques in terms of intraoperative stability and perioperative management requirements.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years.
* American Society of Anesthesiologists (ASA) classification I-IV.
* Scheduled for femoral neck fracture surgery.
* Provided informed consent to participate in the study.

Exclusion Criteria:

* History of allergy to local anesthetics.
* Presence of coagulopathy or bleeding disorders.
* Mental health disorders impairing consent or cooperation.
* Allergy to medications used in the study protocol.
* Presence of infection at the block site.
* Body mass index (BMI) > 30.
* Preoperative or intraoperative conversion to general anesthesia.
* Pregnant patients.
* Severe spinal deformities preventing regional anesthesia application.
* Refusal to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
State Entropy(SE) | Intraoperative period (baseline, 5, 15, 30, 45, 60, 90, and 120 minutes, and end of surgery [up to 3 hours]
  To measure the depth of anesthesia using the State Entropy (SE) index during surgery. SE reflects cortical EEG activity and ranges from 0 to 91. Lower SE values indicate deeper levels of anesthesia. Measurements will be recorded intraoperatively at baseline and at 5, 15, 30, 45, 60, 90, and 120 minutes, as well as at the end of surgery.
Response Entropy(RE) | Intraoperative period (baseline, 5, 15, 30, 45, 60, 90, and 120 minutes, and end of surgery [up to 3 hours]
  To measure the depth of anesthesia using the Response Entropy (RE) index during surgery. RE reflects combined cortical EEG and facial muscle activity and ranges from 0 to 100. Lower RE values indicate deeper levels of anesthesia. Measurements will be recorded intraoperatively at baseline and at 5, 15, 30, 45, 60, 90, and 120 minutes, as well as at the end of surgery.

SECONDARY OUTCOMES:
Surgical Pleth Index (SPI) | Intraoperative period (baseline, 5, 15, 30, 45, 60, 90, and 120 minutes, and end of surgery [up to 3 hours]
  To assess intraoperative nociception and stress levels using the Surgical Pleth Index (SPI). The SPI reflects autonomic responses to surgical stimuli and ranges from 0 to 100. Higher SPI values indicate higher nociception and stress. Measurements will be
Intraoperative Blood Pressure Changes | Intraoperative period (baseline, 5, 15, 30, 45, 60, 90, and 120 minutes, and end of surgery [up to 3 hours]
  To monitor systolic, diastolic, and mean arterial blood pressure changes during surgery.
Sedative Drug Requirement | Entire surgery duration
  Total amount of sedative medications administered intraoperatively, including propofol and fentanyl. The cumulative dose will be recorded throughout the entire surgery duration (propofol in milligrams; fentanyl in micrograms).
Total Intravenous Fluid Volume | Entire surgery duration
  Total volume of intravenous fluids administered intraoperatively. The cumulative fluid amount will be recorded in milliliters (mL) during the entire surgery duration.

CONTACTS AND LOCATIONS:
Locations (1):
- Healt Science University Bursa Yuksek Ihtisas Research and Education Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will not be shared due to privacy and confidentiality concerns.